CLINICAL TRIAL: NCT02065882
Title: A Prospective, Open-label, Phase I/III Study Investigating Pharmacokinetic Properties of BT524 and Efficacy and Safety of BT524 in the Treatment and Prophylaxis of Bleeding in Patients With Congenital Fibrinogen Deficiency
Brief Title: Pharmacokinetic, Efficacy and Safety of BT524 in Patients With Congenital Fibrinogen Deficiency
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biotest (Industry)
Collaborators: ICON plc (Industry); Phoenix Clinical Research (Other); Accovion GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Biotest 984; 2011-004154-25 (EudraCT Number)
Record Dates: First submitted 2014-02-03; First posted 2014-02-19 (Estimated); Results first posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Congenital Afibrinogenemia; Congenital Hypofibrinogenemia
Keywords: fibrinogen, bleeding,
MeSH Terms: conditions — Afibrinogenemia; Hemorrhage

STUDY DESIGN:
Intervention Model Description: The study was divided into two parts: PK/PD Part I and Efficacy Part II. Patients eligible for PK/PD Part I received a fixed dose of 70 mg BT524 per kilogram body weight (BW) via a single intravenous infusion. Part I was followed by Part II. In Part II, patients received a variable, individually tailored dose of BT524 for on-demand prophylaxis (ODP) and/or on-demand treatment (ODT) in case of bleeding events.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BT524 (Experimental): Part I: A single intravenous infusion of BT524 for assessment of PK/PD of BT524.
  Part II: A single or repetitive intravenous infusion(s) of BT524 for on-demand prophylaxis/on-demand treatment of bleeding events.
  Interventions: Drug: BT524 (Part I); Drug: BT524 (Part II)

INTERVENTIONS:
Drug: BT524 (Part I) — Single intravenous infusion of 70 mg BT524 per kg body weight.
  Other Names: Human Fibrinogen Concentrate
Drug: BT524 (Part II) — Single or repetitive intravenous infusion(s) of BT524, depending on the severity of the disorder, location and extent of the bleeding and patient's clinical condition. Dosage based on individual body weight and fibrinogen level.
  Other Names: Human Fibrinogen Concentrate

SUMMARY:
This was a prospective, open-label, multicenter, phase I/III study investigating the 14-day single-dose pharmacokinetic and pharmacodynamic properties, efficacy and safety of BT524 following intravenous administration in the treatment or prophylaxis of bleeding in patients with congenital afibrinogenemia or severe congenital hypofibrinogenemia.

DETAILED DESCRIPTION:
The study was divided into two parts (Part I and Part II). Part I focused on the primary endpoint of the study, 14-day single-dose pharmacokinetics (PK) and 14-day single-dose pharmacodynamics (PD), as well as the assessment of maximum clot firmness (MCF) as a surrogate parameter for efficacy. Part I of the study was followed by Part II, which evaluated the efficacy and safety of single and repetitive administration of BT524 in patients undergoing on-demand prophylaxis (ODP) and/or on-demand treatment (ODT) for various bleeding events [e.g., elective surgery, spontaneous or post-traumatic major bleeding]. All patients who participated in the PK assessment (Part I) without severe post-administration complications ideally continued treatment with BT524 for ODP and/or ODT in Part II.

ELIGIBILITY:
Inclusion Criteria:

* Known congenital afibrinogenemia or severe congenital hypofibrinogenemia
* Plasma fibrinogen activity ≤ 0.5 g/l and antigen ≤ 0.5 g/l
* Male or female
* Age 0 to 75 years, with the first ten patients will be 18 years or older
* Presumed to be compliant with the study procedures and to terminate the study as scheduled
* Willing and able to be hospitalized for 3 days for the pharmacokinetic assessment (if applicable)
* Willing and able to be hospitalized - if required - in case of interventions (e.g., surgical procedures, major bleeds)
* Written informed consent by the patient, his/her parents or by the patient's legal/authorized representative as applicable

Exclusion Criteria:

* Known congenital dysfibrinogenemia (not applicable for adult patients with hypodysfibrinogenemia in study part II)
* Known bleeding disorder other than congenital fibrinogen deficiency
* History of esophageal variceal bleeding
* Known presence or history of venous/arterial thrombosis or thromboembolic event in the preceding 6 months
* Known presence or history of fibrinogen inhibitory antibodies
* Known presence or history of hypersensitivity to human fibrinogen or human plasma proteins e.g., immunoglobulins, vaccines or hypersensitivity to any of the excipients
* Known positive serology for HIV-1 and HIV-2
* Clinically relevant biochemical or hematological findings (except due to underlying disease or emergency bleeding) outside the normal range (at the investigator's discretion)
* Clinically relevant pathological findings in physical examination including electrocardiogram
* Treatment with any fibrinogen concentrate and/or fibrinogen-containing product within 2 weeks prior to infusion of BT524
* Concomitant medication interacting relevantly with the coagulation system such as: low molecular weight heparin or unfractioned heparin, factor Xa inhibitors, thrombin inhibitors (factor II a inhibitors), antiplatelet drugs (PY12 inhibitors) within 2 weeks prior to infusion of BT524
* Recent vaccination (within 3 weeks prior to infusion)
* Body weight (BW) below 22 kg for patients ≥ 6 years; BW below the 5th percentile of the normal range for children < 6 years (refers to local standards)
* End stage disease
* Abuse of drugs
* Unable to understand and follow the study requirements
* Participation in another interventional clinical study within 30 days before entering the study or during the study
* Pregnant/ nursing woman, or woman of childbearing potential not using reliable/ effective contraceptive method(s) during the study and at least one month after the last administration of study drug (e.g., oral/ injectable/ implantable/ insertable/ topical hormonal contraceptives, intrauterine devices, female sterilization, partner's vasectomy or condoms)
* Any other condition that, to the investigator's judgment, could have an impact on patient's safety or the study results
* Elective surgery during the 14 day PK blood sampling period
* Acute infection
* Clinically relevant increase or decrease in body temperature
* Actively bleeding or anticipated bleeding (including female menorrhea) at the time point of or within 7 days prior to infusion of BT524
* Surgery within 7 days prior to infusion of BT524
* Immobilization within 7 days prior to infusion of BT524
* Intake of alcohol or significantly increased intake of caffeine containing products within 24 hours prior to infusion of BT524
* Blood donation or comparable blood loss within 60 days prior to infusion of BT524
* Excessive physical exercise (extreme sports activities, sauna) within 72 hours prior to infusion of BT524

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2020-05-18 (Actual); Study Completion 2020-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Djambas Khayat, MD, Principal Investigator — Hôtel Dieu de France, Dept. of Pediatrics
Locations (6):
- Site 15, Sofia, Bulgaria
- Site 11, Cairo, Egypt
- Site 16, Frankfurt, Germany
- Site 01, Beirut, Lebanon
- Tunisia (2):
  - Site 14, Sousse
  - Site12, Tunis

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Part I and Part II of the study were conducted consecutively, enrolling a total of 67 participants. The total number of participants enrolled (N=67) is smaller than the sum of participants enrolled in Part I (N=35) and Part II (N=59), because 27 participants who successfully completed Part I were subsequently enrolled in Part II. Of the enrolled participants, N=27 in Part I and N=36 in Part II were treated with BT524, with 18 participants receiving BT524 in both parts of the study.
Groups:
- BT542 (Human Fibrinogen Concentrate): Part I: A single intravenous infusion of 70 mg BT524 per kg of body weight.
  Part II: Single or repetitive intravenous infusion(s) of BT524, as individually required.
Period: Part I: PK/PD
Arm/Group | BT542 (Human Fibrinogen Concentrate)
Started | 35
Treated | 27
Completed | 27
Not Completed | 8
Not completed — Screening failure | 5
Not completed — Withdrawal by Subject | 2
Not completed — Adverse Event | 1
Period: Part II: Clinical Efficacy
Arm/Group | BT542 (Human Fibrinogen Concentrate)
Started | 59 (The 27 participants who completed part I successfully were also enrolled in part II. In addition, 32 new participants who had not participated in Part I of the study were enrolled directly into Part II. In total, 59 participants started Part II of the study.)
Treated | 36
Completed | 28
Not Completed | 31
Not completed — Screening failure | 7
Not completed — Withdrawal by Subject | 2
Not completed — Adverse Event | 5
Not completed — Regulatory Authority Decision | 3
Not completed — No Bleeding Event | 11
Not completed — Protocol Violation | 3

BASELINE CHARACTERISTICS:
Population: Part I: Baseline characteristics were assessed in all participants who received any portion of BT524 (n=27).
  Part II: Baseline characteristics were assessed in all participants who received any portion of BT524 (n=36).
Groups:
- BT524 (Human Fibrinogen Concentrate): Part I: A single intravenous infusion of BT524 for assessment of PK/PD of BT524.
  Part II: A single or repetitive intravenous infusion(s) of BT524 for on-demand prophylaxis/on-demand treatment of bleeding events.
Arm/Group | BT524 (Human Fibrinogen Concentrate)
Number analyzed (Participants) | 67
Age, Categorical [Count of Participants; unit: Participants] — Population: Part I: All participants treated with BT524, n=27. Part II: All participants treated with BT524, n=36.
  Participants
    Part I: number analyzed (Participants) | 27
    Part I: <=18 years | 12
    Part I: Between 18 and 65 years | 15
    Part I: >=65 years | 0
    Part II: number analyzed (Participants) | 36
    Part II: <=18 years | 16
    Part II: Between 18 and 65 years | 20
    Part II: >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Part I: All participants treated with BT524, n=27. Part II: All participants treated with BT524, n=36.
  years
    Part I: number analyzed (Participants) | 27
    Part I | 17.6 (11.82)
    Part II: number analyzed (Participants) | 36
    Part II | 19.6 (11.76)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Part I: All participants treated with BT524, n=27. Part II: All participants treated with BT524, n=36.
  Participants
    Part I: number analyzed (Participants) | 27
    Part I: Female | 13
    Part I: Male | 14
    Part II: number analyzed (Participants) | 36
    Part II: Female | 14
    Part II: Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Part I: All participants treated with BT524, n=27. Part II: All participants treated with BT524, n=36.
  Participants
    Part I: number analyzed (Participants) | 27
    Part I: Hispanic or Latino | 0
    Part I: Not Hispanic or Latino | 27
    Part I: Unknown or Not Reported | 0
    Part II: number analyzed (Participants) | 36
    Part II: Hispanic or Latino | 0
    Part II: Not Hispanic or Latino | 36
    Part II: Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Part I: All participants treated with BT524, n=27. Part II: All participants treated with BT524, n=36.
  Participants
    Part I: number analyzed (Participants) | 27
    Part I: American Indian or Alaska Native | 0
    Part I: Asian | 0
    Part I: Native Hawaiian or Other Pacific Islander | 0
    Part I: Black or African American | 1
    Part I: White | 26
    Part I: More than one race | 0
    Part I: Unknown or Not Reported | 0
    Part II: number analyzed (Participants) | 36
    Part II: American Indian or Alaska Native | 0
    Part II: Asian | 0
    Part II: Native Hawaiian or Other Pacific Islander | 0
    Part II: Black or African American | 0
    Part II: White | 36
    Part II: More than one race | 0
    Part II: Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Lebanon | 39
  Egypt | 12
  Bulgaria | 2
  Tunisia | 13
  Germany | 1
Maximum Clot Firmness [Mean (Standard Deviation); unit: mm] — Population: Part I: All particpiants treated with BT524, n=27; MCF values were available for 22 participants. Data were missing for 5 participants: 3 adults, 1 adolescent, 1 child (aged 6 to <12 y). Part II: All participants treated with BT524, n=36.
  mm
    Part I: Adults: number analyzed (Participants) | 12
    Part I: Adults | 1.2 (0.58)
    Part I: Adolescents, 12 to <18 years: number analyzed (Participants) | 2
    Part I: Adolescents, 12 to <18 years | 1.0 (0)
    Part I: Children, 6 to <12 years: number analyzed (Participants) | 2
    Part I: Children, 6 to <12 years | 1.0 (0)
    Part I: Children, <6 years: number analyzed (Participants) | 6
    Part I: Children, <6 years | 1.0 (0)
    Part II: Adults: number analyzed (Participants) | 20
    Part II: Adults | 2.1 (4.03)
    Part II: Adolescents, 12 to <18 years: number analyzed (Participants) | 4
    Part II: Adolescents, 12 to <18 years | 1.0 (0)
    Part II: Children, 6 to <12 years: number analyzed (Participants) | 9
    Part II: Children, 6 to <12 years | 1.0 (0)
    Part II: Children, <6 years: number analyzed (Participants) | 3
    Part II: Children, <6 years | 1.0 (0)
Fibrinogen Activity [Mean (Standard Deviation); unit: g/L] — Population: Part I: All participants treated with BT524, n=27. Part II: All participants treated with BT524, n=36. Fibrinogen Activity was measured in all participants prior to BT524 treatment.
  g/L
    Part I: Adults: number analyzed (Participants) | 15
    Part I: Adults | 0.1750 (0)
    Part I: Adolescents, 12 to <18 years: number analyzed (Participants) | 3
    Part I: Adolescents, 12 to <18 years | 0.1750 (0)
    Part I: Children, 6 to <12 years: number analyzed (Participants) | 3
    Part I: Children, 6 to <12 years | 0.1750 (0)
    Part I: Children, <6 years: number analyzed (Participants) | 6
    Part I: Children, <6 years | 0.1500 (0)
    Part II: Adults: number analyzed (Participants) | 20
    Part II: Adults | 0.1681 (0.01856)
    Part II: Adolescents, 12 to <18 years: number analyzed (Participants) | 4
    Part II: Adolescents, 12 to <18 years | 0.1578 (0.01611)
    Part II: Children, 6 to <12 years: number analyzed (Participants) | 9
    Part II: Children, 6 to <12 years | 0.1553 (0.02385)
    Part II: Children, <6 years: number analyzed (Participants) | 3
    Part II: Children, <6 years | 0.1500 (0)
Disease characteristics [Count of Participants; unit: Participants] — Population: Part I: All participants treated with BT524, n=27. Part II: All participants treated with BT524, n=36.
  Participants
    Part I: number analyzed (Participants) | 27
    Part I: Afibrinogenemia | 27
    Part I: Severe Hypofibrinogenemia | 0
    Part II: number analyzed (Participants) | 36
    Part II: Afibrinogenemia | 34
    Part II: Severe Hypofibrinogenemia | 2

OUTCOME MEASURES:

1. Primary Outcome: Single-dose Pharmacokinetics (PK) of BT524: Terminal Elimination Half-life (t1/2) for Fibrinogen Antigen
Description: T1/2 of fibrinogen antigen was determined from samples taken at several time points during the 14 day sampling period. T1/2 was derived from time-concentration profiles using adapted methodology (non-compartmental analysis, compartment analysis, or population modeling, as appropriate/ required).
Time Frame: Pre-dose on Dosing Day 0, at the end of the infusion and 0.5, 1, 2, 4, 8, 24, 48, 96, 168, 240 and 336 hours post-dose
Population: PK Set: consists of all patients of part I with PK data.
Measure: Mean (Standard Deviation); unit: hours
Groups:
- BT524 (Human Fibrinogen Concentrate): Part I: A single intravenous infusion of 70 mg BT524 per kg body weight for assessment of PK/PD of BT524.
Arm/Group | BT524 (Human Fibrinogen Concentrate)
Number analyzed (Participants) | 27
hours | 67.9 (15.3)

2. Primary Outcome: Single-dose Pharmacokinetics (PK) of BT524: Time to Maximum Concentration (Tmax) for Fibrinogen Antigen
Description: Time of occurence of Cmax relative to dosing (Tmax) for fibrinogen antigen was determined from samples taken at several time points during the 14 day sampling period. Tmax was derived from time-concentration profiles using adapted methodology (non-compartmental analysis, compartment analysis, or population modeling, as appropriate/required).
Time Frame: Pre-dose on Dosing Day 0, at the end of the infusion and 0.5, 1, 2, 4, 8, 24, 48, 96, 168, 240 and 336 hours post-dose
Population: PK Set: consists of all patients of part I with PK data.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | BT524 (Human Fibrinogen Concentrate)
Number analyzed (Participants) | 27
hours | 0.843 (0.361)

3. Primary Outcome: Single-Dose Pharmacokinetics (PK) for BT524: Maximum Concentration (Cmax) for Fibrinogen Antigen
Description: Maximum observed plasma concentration (Cmax) for fibrinogen antigen was determined from samples taken at several time points during the 14 day sampling period. Cmax was derived from time-concentration profiles using adapted methodology (non-compartmental analysis, compartment analysis, or population modeling, as appropriate/ required).
Time Frame: Pre-dose on Dosing Day 0, at the end of the infusion and 0.5, 1, 2, 4, 8, 24, 48, 96, 168, 240 and 336 hours post-dose
Population: PK Set: consists of all patients of part I with PK data.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | BT524 (Human Fibrinogen Concentrate)
Number analyzed (Participants) | 27
g/L | 1.81 (0.423)

4. Primary Outcome: Single-Dose Pharmacokinetics (PK) for BT524: Area Under the Curve (AUC) Calculated to the Last Measured Concentration (AUC0-tz) for Fibrinogen Antigen
Description: AUC0-tz: Area under the time course of the plasma concentrations calculated from time zero up to the last quantifiable plasma concentration for fibrinogen antigen, was determined from samples taken at several time points during the 14 day sampling period. AUC0-tz was derived from time-concentration profiles using adapted methodology (noncompartmental analysis, compartment analysis, or population modeling, as appropriate/ required).
Time Frame: Pre-dose on Dosing Day 0, at the end of the infusion and 0.5, 1, 2, 4, 8, 24, 48, 96, 168, 240 and 336 hours post-dose
Population: PK Set: consists of all patients of part I with PK data.
Measure: Mean (Standard Deviation); unit: g*h/L
Arm/Group | BT524 (Human Fibrinogen Concentrate)
Number analyzed (Participants) | 27
g*h/L | 144 (38.9)

5. Primary Outcome: Single-Dose Pharmacokinetics (PK) for BT524: Extent of Area Under the Curve (AUC) Extrapolation Beyond Last Concentration (AUCextr) for Fibrinogen Antigen
Description: AUCextr: extent of AUC extrapolation beyond last concentration for fibrinogen antigen, was determined from samples taken at several time points during the 14 day sampling period. AUCextr was derived from time-concentration profiles using adapted methodology (non-compartmental analysis, compartment analysis, or population modeling, as appropriate/ required).
Time Frame: Pre-dose on Dosing Day 0, at the end of the infusion and 0.5, 1, 2, 4, 8, 24, 48, 96, 168, 240 and 336 hours post-dose
Population: PK Set: consists of all patients of part I with PK data.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | BT524 (Human Fibrinogen Concentrate)
Number analyzed (Participants) | 27
percentage | 17.1 (3.58)

6. Primary Outcome: Single-Dose Pharmacokinetics (PK) for BT524: Area Under the Curve (AUC) From Time 0 to Infinity (AUC0-∞) for Fibrinogen Antigen
Description: AUC0-∞: AUC from time 0 to infinity for fibrinogen antigen, was determined from samples taken at several time points during the 14 day sampling period. AUC0-∞ was derived from time-concentration profiles using adapted methodology (non-compartmental analysis, compartment analysis, or population modeling, as appropriate/ required).
Time Frame: Pre-dose on Dosing Day 0, at the end of the infusion and 0.5, 1, 2, 4, 8, 24, 48, 96, 168, 240 and 336 hours post-dose
Population: PK Set: consists of all patients of part I with PK data.
Measure: Mean (Standard Deviation); unit: g*h/L
Arm/Group | BT524 (Human Fibrinogen Concentrate)
Number analyzed (Participants) | 27
g*h/L | 173 (45.4)

7. Primary Outcome: Single-Dose Pharmacokinetics (PK) for BT524: Mean Residence Time (MRT) Extrapolated to Infinity (MRT0-∞) for Fibrinogen Antigen
Description: MRT0-∞: Mean Residence Time (MRT) extrapolated to infinity for fibrinogen antigen was determined from samples taken at several time points during the 14 day sampling period. MRT0-∞ was derived from time-concentration profiles using adapted methodology (non-compartmental analysis, compartment analysis, or population modeling, as appropriate/ required).
Time Frame: Pre-dose on Dosing Day 0, at the end of the infusion and 0.5, 1, 2, 4, 8, 24, 48, 96, 168, 240 and 336 hours post-dose
Population: PK Set: consists of all patients of part I with PK data.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | BT524 (Human Fibrinogen Concentrate)
Number analyzed (Participants) | 27
hours | 133 (17.4)

8. Primary Outcome: Single-Dose Pharmacokinetics (PK) for BT524: Clearance (CL) for Fibrinogen Antigen
Description: CL: Total clearance (CL) for fibrinogen antigen was determined from samples taken at several time points during the 14 day sampling period. CL was derived from time-concentration profiles using adapted methodology (non-compartmental analysis, compartment analysis, or population modeling, as appropriate/ required).
Time Frame: Pre-dose on Dosing Day 0, at the end of the infusion and 0.5, 1, 2, 4, 8, 24, 48, 96, 168, 240 and 336 hours post-dose
Population: PK Set: consists of all patients of part I with PK data.
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | BT524 (Human Fibrinogen Concentrate)
Number analyzed (Participants) | 27
L/h | 0.0206 (0.00961)

9. Primary Outcome: Single-Dose Pharmacokinetics (PK) for BT524: Volume of Distribution at Presumed Steady-state (Vdss) for Fibrinogen Antigen
Description: Vdss: Volume of distribution at presumed steady-state for fibrinogen antigen was determined from samples taken at several time points during the 14 day sampling period. Vdss was derived from time-concentration profiles using adapted methodology (non-compartmental analysis, compartment analysis, or population modeling, as appropriate/ required).
Time Frame: Pre-dose on Dosing Day 0, at the end of the infusion and 0.5, 1, 2, 4, 8, 24, 48, 96, 168, 240 and 336 hours post-dose
Population: PK Set: consists of all patients of part I with PK data.
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | BT524 (Human Fibrinogen Concentrate)
Number analyzed (Participants) | 27
Liter | 2.70 (1.34)

10. Primary Outcome: Single-Dose Pharmacokinetics (PK) for BT524: Volume of Distribution at Presumed Steady-state (Vdss) Per kg Body Weight (BW) for Fibrinogen Antigen
Description: Vdss per kg BW: Volume of distribution at presumed steady-state per kg bodyweight for fibrinogen antigen was determined from samples taken at several time points during the 14 day sampling period. Vdss per kg BW was derived from time-concentration profiles using adapted methodology (non-compartmental analysis, compartment analysis, or population modeling, as appropriate/ required).
Time Frame: Pre-dose on Dosing Day 0, at the end of the infusion and 0.5, 1, 2, 4, 8, 24, 48, 96, 168, 240 and 336 hours post-dose
Population: PK Set: consists of all patients of part I with PK data.
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | BT524 (Human Fibrinogen Concentrate)
Number analyzed (Participants) | 27
mL/kg | 57.8 (19.1)

11. Primary Outcome: Single-Dose Pharmacokinetics (PK) for BT524: Incremental Recovery (IR) for Fibrinogen Antigen
Description: IR is the dose-adjusted maximum fibrinogen increase in plasma within 4 hours after the end of infusion.
Time Frame: Between pre-dose and 4 hours post-dose
Population: PK Set: consists of all patients of part I with PK data.
Measure: Mean (Standard Deviation); unit: (mg/dL)/(mg/kg dose)
Arm/Group | BT524 (Human Fibrinogen Concentrate)
Number analyzed (Participants) | 27
(mg/dL)/(mg/kg dose) | 2.63 (0.652)

12. Primary Outcome: Single-Dose Pharmacokinetics (PK) for BT524: Classical in Vivo Recovery (CIR) for Fibrinogen Antigen
Description: CIR: maximum fibrinogen increase in plasma within 4 hours after the end of infusion divided by the maximum theoretical fibrinogen increase
Time Frame: Between pre-dose and 4 hours post-dose
Population: PK Set: consists of all patients of part I with PK data.
Measure: Mean (Standard Deviation); unit: % of expected increase in fibrinogen
Arm/Group | BT524 (Human Fibrinogen Concentrate)
Number analyzed (Participants) | 27
% of expected increase in fibrinogen | 118 (29.4)

13. Secondary Outcome: Single-dose Pharmacodynamics (PD) of BT524: Terminal Elimination Half-life (t1/2) for Fibrinogen Activity
Description: T1/2 of fibrinogen activity was determined from samples taken at several time points during the 14 day sampling period. T1/2 was derived from time-concentration profiles using adapted methodology (non-compartmental analysis, compartment analysis, or population modeling, as appropriate/ required).
Time Frame: Pre-dose on Dosing Day 0, at the end of the infusion and 0.5, 1, 2, 4, 8, 24, 48, 96, 168, 240 and 336 hours post-dose
Population: PK Set: consists of all patients of part I with PK data.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | BT524 (Human Fibrinogen Concentrate)
Number analyzed (Participants) | 27
hours | 60.3 (13.3)

14. Secondary Outcome: Single-dose Pharmacodynamics (PD) of BT524: Time to Maximum Concentration (Tmax) for Fibrinogen Activity
Description: Time of occurence of Cmax relative to dosing (Tmax) for fibrinogen activity was determined from samples taken at several time points during the 14 day sampling period. Tmax was derived from time-concentration profiles using adapted methodology (non-compartmental analysis, compartment analysis, or population modeling, as appropriate/required).
Time Frame: Pre-dose on Dosing Day 0, at the end of the infusion and 0.5, 1, 2, 4, 8, 24, 48, 96, 168, 240 and 336 hours post-dose
Population: PK Set: consists of all patients of part I with PK data.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | BT524 (Human Fibrinogen Concentrate)
Number analyzed (Participants) | 27
hours | 0.843 (0.361)

15. Secondary Outcome: Single-dose Pharmacodynamics (PD) of BT524: Maximum Concentration (Cmax) for Fibrinogen Activity
Description: Maximum observed plasma concentration (Cmax) for fibrinogen activity was determined from samples taken at several time points during the 14 day sampling period. Cmax was derived from time-concentration profiles using adapted methodology (non-compartmental analysis, compartment analysis, or population modeling, as appropriate/ required).
Time Frame: Pre-dose on Dosing Day 0, at the end of the infusion and 0.5, 1, 2, 4, 8, 24, 48, 96, 168, 240 and 336 hours post-dose
Population: PK Set: consists of all patients of part I with PK data.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | BT524 (Human Fibrinogen Concentrate)
Number analyzed (Participants) | 27
g/L | 1.26 (0,396)

16. Secondary Outcome: Single-dose Pharmacodynamics (PD) of BT524: Area Under the Curve (AUC) Calculated to the Last Measured Concentration (AUC0-tz) for Fibrinogen Activity
Description: AUC0-tz: Area under the time course of the plasma concentrations calculated from time zero up to the last quantifiable plasma concentration for fibrinogen activity, was determined from samples taken at several time points during the 14 day sampling period. AUC0-tz was derived from time-concentration profiles using adapted methodology (noncompartmental analysis, compartment analysis, or population modeling, as appropriate/ required).
Time Frame: Pre-dose on Dosing Day 0, at the end of the infusion and 0.5, 1, 2, 4, 8, 24, 48, 96, 168, 240 and 336 hours post-dose
Population: PK Set: consists of all patients of part I with PK data.
Measure: Mean (Standard Deviation); unit: g*h/L
Arm/Group | BT524 (Human Fibrinogen Concentrate)
Number analyzed (Participants) | 27
g*h/L | 88.2 (29.3)

17. Secondary Outcome: Single-dose Pharmacodynamics (PD) of BT524: Extent of Area Under the Curve (AUC) Extrapolation Beyond Last Concentration (AUCextr) for Fibrinogen Activity
Description: AUCextr: extent of AUC extrapolation beyond last concentration for fibrinogen activity, was determined from samples taken at several time points during the 14 day sampling period. AUCextr was derived from time-concentration profiles using adapted methodology (non-compartmental analysis, compartment analysis, or population modeling, as appropriate/ required).
Time Frame: Pre-dose on Dosing Day 0, at the end of the infusion and 0.5, 1, 2, 4, 8, 24, 48, 96, 168, 240 and 336 hours post-dose
Population: PK Set: consists of all patients of part I with PK data.
Measure: Mean (Standard Deviation); unit: percentage (extent of AUC extrapolation)
Arm/Group | BT524 (Human Fibrinogen Concentrate)
Number analyzed (Participants) | 27
percentage (extent of AUC extrapolation) | 15.4 (3.41)

18. Secondary Outcome: Single-dose Pharmacodynamics (PD) of BT524: Area Under the Curve (AUC) From Time 0 to Infinity (AUC0-∞) for Fibrinogen Activity
Description: AUC0-∞: AUC from time 0 to infinity for fibrinogen activity, was determined from samples taken at several time points during the 14 day sampling period. AUC0-∞ was derived from time-concentration profiles using adapted methodology (non-compartmental analysis, compartment analysis, or population modeling, as appropriate/ required).
Time Frame: Pre-dose on Dosing Day 0, at the end of the infusion and 0.5, 1, 2, 4, 8, 24, 48, 96, 168, 240 and 336 hours post-dose
Population: PK Set: consists of all patients of part I with PK data.
Measure: Mean (Standard Deviation); unit: g*h/L
Arm/Group | BT524 (Human Fibrinogen Concentrate)
Number analyzed (Participants) | 27
g*h/L | 104 (33.5)

19. Secondary Outcome: Single-dose Pharmacodynamics (PD) of BT524: Mean Residence Time (MRT) Extrapolated to Infinity (MRT0-∞) for Fibrinogen Activity
Description: MRT0-∞: Mean Residence Time (MRT) extrapolated to infinity for fibrinogen activity was determined from samples taken at several time points during the 14 day sampling period. MRT0-∞ was derived from time-concentration profiles using adapted methodology (non-compartmental analysis, compartment analysis, or population modeling, as appropriate/ required).
Time Frame: Pre-dose on Dosing Day 0, at the end of the infusion and 0.5, 1, 2, 4, 8, 24, 48, 96, 168, 240 and 336 hours post-dose
Population: PK Set: consists of all patients of part I with PK data.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | BT524 (Human Fibrinogen Concentrate)
Number analyzed (Participants) | 27
hours | 124 (16.2)

20. Secondary Outcome: Single-Dose Pharmacodynamics (PD) for BT524: Clearance (CL) for Fibrinogen Activity
Description: CL: Total clearance (CL) for fibrinogen activity was determined from samples taken at several time points during the 14 day sampling period. CL was derived from time-concentration profiles using adapted methodology (non-compartmental analysis, compartment analysis, or population modeling, as appropriate/ required).
Time Frame: Pre-dose on Dosing Day 0, at the end of the infusion and 0.5, 1, 2, 4, 8, 24, 48, 96, 168, 240 and 336 hours post-dose
Population: PK Set: consists of all patients of part I with PK data.
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | BT524 (Human Fibrinogen Concentrate)
Number analyzed (Participants) | 27
L/h | 0.0351 (0.0179)

21. Secondary Outcome: Single-Dose Pharmacodynamics (PD) for BT524: Volume of Distribution at Presumed Steady-state (Vdss) for Fibrinogen Activity
Description: Vdss: Volume of distribution at presumed steady-state for fibrinogen activity was determined from samples taken at several time points during the 14 day sampling period. Vdss was derived from time-concentration profiles using adapted methodology (non-compartmental analysis, compartment analysis, or population modeling, as appropriate/ required).
Time Frame: Pre-dose on Dosing Day 0, at the end of the infusion and 0.5, 1, 2, 4, 8, 24, 48, 96, 168, 240 and 336 hours post-dose
Population: PK Set: consists of all patients of part I with PK data.
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | BT524 (Human Fibrinogen Concentrate)
Number analyzed (Participants) | 27
Liter | 4.31 (2.36)

22. Secondary Outcome: Single-Dose Pharmacodynamics (PD) for BT524: Volume of Distribution at Presumed Steady-state (Vdss) Per kg Body Weight (BW) for Fibrinogen Activity
Description: Vdss per kg BW: Volume of distribution at presumed steady-state per kg bodyweight for fibrinogen activity was determined from samples taken at several time points during the 14 day sampling period. Vdss per kg BW was derived from time-concentration profiles using adapted methodology (non-compartmental analysis, compartment analysis, or population modeling, as appropriate/ required).
Time Frame: Pre-dose on Dosing Day 0, at the end of the infusion and 0.5, 1, 2, 4, 8, 24, 48, 96, 168, 240 and 336 hours post-dose
Population: PK Set: consists of all patients of part I with PK data.
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | BT524 (Human Fibrinogen Concentrate)
Number analyzed (Participants) | 27
mL/kg | 92.4 (34.7)

23. Secondary Outcome: Single-Dose Pharmacodynamics (PD) for BT524: Incremental Recovery (IR) for Fibrinogen Activity
Description: IR is the dose-adjusted maximum fibrinogen increase in plasma within 4 hours after the end of infusion.
Time Frame: Between pre-dose and 4 hours post-dose
Population: PK Set: consists of all patients of part I with PK data.
Measure: Mean (Standard Deviation); unit: (mg/dL)/(mg/kg dose)
Arm/Group | BT524 (Human Fibrinogen Concentrate)
Number analyzed (Participants) | 27
(mg/dL)/(mg/kg dose) | 1.88 (0.610)

24. Secondary Outcome: Single-Dose Pharmacodynamics (PD) for BT524: Classical in Vivo Recovery (CIR) for Fibrinogen Activity
Description: as for outcome 12
Time Frame: Between pre-dose and 4 hours post-dose
Population: PK Set: consists of all patients of part I with PK data.
Measure: Mean (Standard Deviation); unit: % of expected increase in fibrinogen
Arm/Group | BT524 (Human Fibrinogen Concentrate)
Number analyzed (Participants) | 27
% of expected increase in fibrinogen | 84.8 (27.5)

25. Secondary Outcome: Change in Maximum Clot Firmness at 1 Hour Post-end of Infusion
Description: Maximum Clot Firmness (MCF), assessed by rotational thromboelastometry (ROTEM), was used as a surrogate marker of haemostatic efficacy following administration of BT524. In Part I, MCF was measured before and 1 hour after the end of a single BT524 infusion. In Part II, MCF was measured before and 1 hour after the end of each BT524 infusion administered to treat bleeding events. The variable was the change in MCF from pre-dose to 1 hour post-end of infusion.
Time Frame: Part I: pre-dose and at 1 hour post-end of infusion. Part II: pre-dose and at 1 hour post-end of infusion of each bleeding event.
Population: Full analysis set (FAS I/II): all patients who received any portion of BT524 and had at least one efficacy assessment in part I/part II
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: BT524 infusion
Groups:
- Part I: A single intravenous infusion of BT524 for assessment of PK/PD of BT524.
- Part II: A single or repetitive intravenous infusion(s) of BT524 for on-demand prophylaxis/on-demand treatment of bleeding events.
Arm/Group | Part I | Part II
Number analyzed (Participants) | 19 | 36
Number analyzed (BT524 infusion) | 19 | 128
mm
  Adults: number analyzed (Participants) | 12 | 20
  Adults: number analyzed (BT524 infusion) | 12 | 56
  Adults | 11.1 (5.07) | 11.1 (5.55)
  Adolescents, 12 to <18 years: number analyzed (Participants) | 2 | 4
  Adolescents, 12 to <18 years: number analyzed (BT524 infusion) | 2 | 26
  Adolescents, 12 to <18 years | 11.0 (2.83) | 9.8 (5.28)
  Children, 6 to <12 years: number analyzed (Participants) | 2 | 9
  Children, 6 to <12 years: number analyzed (BT524 infusion) | 2 | 43
  Children, 6 to <12 years | 16.5 (3.54) | 11.1 (4.57)
  Children, <6 years: number analyzed (Participants) | 3 | 3
  Children, <6 years: number analyzed (BT524 infusion) | 3 | 3
  Children, <6 years | 9.3 (1.53) | 8.7 (5.51)
Statistical Analysis 1: Comparison: Part I; Test type: Other — Confirmatory t-test testing of the MCF difference (1 h post-dose minus pre-dose); p < 0.0001, t-test, 2 sided

26. Secondary Outcome: Clinical Efficacy for BT524: Overall Hemostatic Response to Treatment With BT524 in Study Part II
Description: Overall hemostatic response (OHR) to treatment with BT524 for each surgical procedure and each treated bleed was rated on a 4-point scale ("none", "moderate", "good" or "excellent"). The sum of good and excellent ratings was defined as "success" in the analysis. Frequencies and percentages of OHR on event level (Success rate in % = number of successfully treated bleeding events / total number of bleeding events).
Time Frame: Part II: Up to 24 hours after end of infusion, or on day of hospital discharge (if between 24 hours and 49 days post-infusion); at the latest on day 49 after the treated bleeding event.
Population: Full bleeding event set (FBE): All bleeding events treated with any portion of BT524 and with at least one efficacy assessment during part II of the study.
Measure: Count of Units; unit: Bleeding Events
Units Other Than Participants: Bleeding Events
Arm/Group | Part II
Number analyzed (Participants) | 36
Number analyzed (Bleeding Events) | 175
Bleeding Events
  Excellent | 150
  Good | 23
  Moderate | 2
  None | 0

27. Secondary Outcome: Clinical Efficacy for BT524: Total Loss of Blood for Surgical Bleeding Events in Study Part II
Description: Total loss of blood was rated by the investigator per surgical bleeding events (eg, intra- and post-operatively, rebleedings) using the classifications of "lower than expected", "within the expected range", and "higher than expected". The ratings were analyzed descriptively (frequencies and percentages) on event level for the Full Bleeding Event Set (FBE).
Time Frame: as for outcome 26
Population: as for outcome 26
Measure: Count of Units; unit: Surgical bleeding events
Units Other Than Participants: Surgical bleeding events
Arm/Group | Part II
Number analyzed (Participants) | 36
Number analyzed (Surgical bleeding events) | 54
Surgical bleeding events
  Loss of blood is lower than expected for the procedure performed. | 3
  Loss of blood is within the expected range for the procedure performed. | 45
  Loss of blood is higher than expected for the procedure performed. | 4
  Missing | 2

28. Secondary Outcome: Clinical Efficacy for BT524: Units of Other Fibrinogen-containing Products (FCP) Infused Besides BT524 in Study Part II
Description: Units of other fibrinogen-containing products (FCP) infused besides BT524 eg, fresh frozen plasma (FFP) or cryoprecipitate or alternative commercially available fibrinogen concentrates given to counteract hemodynamic instability were documented and analyzed descriptively on event level for the FBE.
Time Frame: as for outcome 26
Population: as for outcome 26
Measure: Number; unit: Number of FCP
Units Other Than Participants: Bleeding Events
Arm/Group | Part II
Number analyzed (Participants) | 36
Number analyzed (Bleeding Events) | 175
Number of FCP | 0

ADVERSE EVENTS:
Time Frame: Day 0 to Day 49 (From the day of study drug administration until 49±4 days after the last administration of the study drug in Part I, up to 1 year in Part II.
Description: Adverse Events (AEs) reported from the time of study drug administration to the safety visit on Day 49± 4 were recorded as treatment-emergent adverse events (TEAEs).
Groups:
- PK/PD Part I: Part I: A single intravenous infusion of 70 mg BT524 per kg body weight for assessment of PK/PD of BT524.
- Part II: Part II: A single or repetitive intravenous infusion(s) of BT524 as individually required, for on-demand prophylaxis/on-demand treatment of bleeding events.
Arm/Group | PK/PD Part I | Part II
All-Cause Mortality (participants affected / at risk) | 0/27 | 1/36
Serious Adverse Events (participants affected / at risk) | 2/27 | 7/36
Other Adverse Events (participants affected / at risk) | 10/27 | 25/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PK/PD Part I (N=27) | Part II (N=36)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Extradural heamatoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Hypertensive encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Post streptococcal glomerulonephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PK/PD Part I (N=27) | Part II (N=36)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 2 (3)
Toothache (Gastrointestinal disorders) | 2 (2) | 3 (3)
Pyrexia (General disorders) | 1 (1) | 3 (3)
Swelling face (General disorders) | 0 (0) | 3 (3)
Rhinitis (Infections and infestations) | 1 (1) | 2 (2)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 9 (30)
Skin wound (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 (1) | 6 (10)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 4 (5)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Osteorrhagia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (9)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (8)
Headache (Nervous system disorders) | 1 (1) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Haematoma (Vascular disorders) | 0 (0) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (3):
  • Study Protocol (2018-05-08): https://cdn.clinicaltrials.gov/large-docs/82/NCT02065882/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-02): https://cdn.clinicaltrials.gov/large-docs/82/NCT02065882/SAP_001.pdf
  • Informed Consent Form (2018-08-02): https://cdn.clinicaltrials.gov/large-docs/82/NCT02065882/ICF_002.pdf